CLINICAL TRIAL: NCT03288766
Title: A Single-Arm Prospective, Multi-Centered Study to Assess the SHERLOCK 3CG™ Diamond Tip Confirmation System
Brief Title: SHERLOCK 3CG™ Diamond Tip Confirmation System
Acronym: MODUS II
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: BAS-14-003
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-01

CONDITIONS: Indication for Peripheral Intravenous Catheterization; Atrial Flutter; Premature Atrial Contraction; Premature Ventricular Contraction; Premature Junctional Contraction; Tachycardia; Atrioventricular Block; Bundle-Branch Block
MeSH Terms: conditions — Atrial Flutter; Atrial Premature Complexes; Ventricular Premature Complexes; Tachycardia; Atrioventricular Block; Bundle-Branch Block | interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PICC Placement with Study Device: PICC Placement with SHERLOCK 3CG™ Diamond TCS with MODUS II software
  Interventions: Procedure: PICC placement with SHERLOCK 3CG™ Diamond TCS with MODUS II software

INTERVENTIONS:
Procedure: PICC placement with SHERLOCK 3CG™ Diamond TCS with MODUS II software — The SHERLOCK 3CG™ Diamond Tip Confirmation System (TCS) is an FDA-cleared fully-integrated magnetic tracking and ECG-based PICC tip confirmation technology, indicated for use as an alternative to chest x-ray and fluoroscopy for PICC tip placement confirmation in adult patients without any alterations of cardiac rhythms that change the normal presentation of the P-wave. A software package, MODUS II, has been developed to accurately analyze the entire ECG complex and identify the correct placement of the PICC tip based on a patient's individual ECG, in the absence of an easily identifiable P-wave. This software system is designed to provide visual and/or audio cues to notify the PICC placer of the location of the PICC tip relative to the cavoatrial junction (CAJ) of the patient.

SUMMARY:
This study is a single-arm, prospective, multi-center study to assess clinical performance of the SHERLOCK 3CG™ Diamond Tip Confirmation System (TCS) with MODUS II software for confirming correct tip position of peripherally inserted central catheters (PICCs) in adult subjects with altered cardiac rhythm.

DETAILED DESCRIPTION:
This study is intended to confirm the accuracy of the SHERLOCK 3CG™ Diamond TCS with the addition of MODUS II (SLM2) software to eliminate the need for post-procedural chest x-ray (CXR) in adult subjects with cardiac abnormalities that alter presentation of the P-wave. Atrial fibrillation will be the primary target while data on pacemaker driven rhythms and other arrhythmia types will also be collected to explore overall performance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 21 years of age with altered cardiac rhythm (no recognizable P-wave on standard ECG) with diagnosis of specific arrhythmia type or identification of pacemaker driven rhythms as defined below:

  1. Atrial fibrillation with history of diagnosis per 12-lead ECG in medical record or diagnosed via bedside telemetry by study team RN at assessment, or
  2. All other arrhythmias (including but not limited to atrial flutter, PAC, PVC, PJC, tachycardia, AV Block, BB Block) with history of diagnosis per 12-lead ECG in medical record or diagnosed via bedside telemetry by cardiac unit RN at assessment, or retrospectively by site cardiologist, or
  3. Pacemaker driven rhythm with temporary or permanent pacemaker device in place;
* Subject requires PICC placement as part of standard of care;
* Subject or Legally Authorized Representative (LAR) has signed an Informed Consent Form (ICF).

Exclusion Criteria:

* Subject has a contraindication to PICC placement as listed in the Instructions for Use (IFU) to include:

  1. The presence of bacteremia or septicemia (known or suspected),
  2. The patient's body size is insufficient to accommodate the size of the implanted device,
  3. The patient is known or is suspected to be allergic to materials contained in the device,
  4. Past irradiation of prospective insertion site,
  5. Previous episodes of venous thrombosis or vascular surgical procedures at the prospective placement site,
  6. Local tissue factors will prevent proper device stabilization and/or access;
* Subjects who previously had a PICC in place and require a PICC exchange;
* Subject has presence of active resting tremor (i.e. Parkinson's, Multiple Sclerosis, etc.) deemed by Investigator to have potential impact on procedure accuracy;
* Subjects who are pregnant or think they may be pregnant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be adult males or females ≥ 21 years of age with identifiable alterations of cardiac rhythm. For this study, altered cardiac rhythm is defined as any condition that does not have a P-wave on ECG.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Rate of successful PICC tip placement within the lower third of the superior vena cava (SVC) or in the cavoatrial junction (CAJ) using SLM2 | The PICC insertion procedure is 60-90 mins in duration
  Tip positioning is determined at bedside by the software via the Green Diamond Indicator (GDI+) and confirmed by CXR. PICC tip placement will be considered successful if it is determined to be in the lower 1/3 of the SVC or in the CAJ by an independent, blinded radiologist judging position retrospectively against pre-specified anatomical criteria.

SECONDARY OUTCOMES:
Rate of successful PICC tip placement within the lower third of the superior vena cava (SVC) or in the cavoatrial junction (CAJ) using SLM2 in the absence of a GDI | The PICC insertion procedure is 60-90 mins in duration
  It is expected there will be some cases where the MODUS II software may fail to present a Green Diamond Indicator (GDI-). In the absence of a GDI, tip positioning is determined at bedside using magnetic tracking and external measurement per hospital protocol, with CXR required for tip confirmation. PICC tip placement will be considered successful if it is determined to be in the lower 1/3 of the SVC or in the CAJ by an independent, blinded radiologist judging position retrospectively against pre-specified anatomical criteria.
Percent agreement between the site readings of the CXR (standard of care) versus those completed by an independent, blinded radiologist | The PICC insertion procedure is 60-90 mins in duration
  An independent, blinded radiologist will judge PICC tip position retrospectively against pre-specified anatomical criteria compared with findings of the SLM2.

CONTACTS AND LOCATIONS:
Overall Officials: Rushil Sankpal, Study Director — Becton Dickinson
Locations (8):
- United States (6):
  - Summerlin Hospital and Medical Center, Las Vegas, Nevada
  - Moses Cone Hospital, Greensboro, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - J.W. Ruby Memorial Hospital, Morgantown, West Virginia
- Australia (2):
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Fiona Stanley Hospital, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: No